CLINICAL TRIAL: NCT06307561
Title: The Effect of Dystonia Severity on Participation in Daily Living Activities and Caregivers in Children of Cerebral Palsy With Secondary Dystonia
Status: Completed | Type: Observational
Sponsor: Acıbadem Atunizade Hospital (Other)
Responsible Party: Principal Investigator, Gizem Gurzoglu, Pediatric Physiotherapist, Acıbadem Atunizade Hospital
Other Study IDs: GGurzoglu
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Secondary Dystonia; Cerebral Palsy, Mixed
Keywords: Dystonia; Participation; Caregiver; Burden
MeSH Terms: conditions — Dystonic Disorders; Cerebral Palsy; Dystonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dystonia is the most common movement disorder in the pediatric population after spasticity. It can affect normal motor development and cause significant motor retardation. The presence of dystonia may affect motor function, pain, and ease of care in CP. Additionally, it can cause serious difficulties in daily living activities and social participation and long-term joint deformity. The increase in the severity of dystonia in CP children with secondary dystonia may affect the quality of life, activity and participation of the children, as well as the caregiver. The importance of caregivers is an undeniable fact, especially in these patient groups. This study aims to investigate the burden of dystonia severity on the participation in daily living activities and caregivers of children with CP with secondary dystonia.

DETAILED DESCRIPTION:
It's an observational study. Purpose of the study: Investigating the burden of dystonia severity on the participation in daily living activities and caregivers of children with CP with secondary dystonia.

* Does dystonia severity affect participation in daily life activities in CP children with secondary dystonia?
* Does the severity of dystonia in children with CP with secondary dystonia affect the burden on the caregiver?
* Are the participation in daily living activities and caregiver burden of children with CP with secondary dystonia related to each other?

Total of 20 CP cases with secondary dystonia who applied to Acıbadem University Department of Pediatric Neurosurgery will be included in the study.

Dystonia severity of these cases will be evaluated with the Barry-Albright Dystonia Scale (BADS). Children's participation in daily living activities will be evaluated with The Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD), and the burden on the caregiver will be evaluated with the Care and Comfort Hypertonicity Questionnaire (CCHQ).

ELIGIBILITY:
Inclusion Criteria:

* Total of 20 cases CP with secondary dystonia, aged between 3-15 years were included in the study.
* Obtaining voluntary consent from the family.

Exclusion Criteria:

* Having a surgical operation procedure on the musculoskeletal system.
* Receiving BoNT-A in the last 6 months.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Total of 20 cases CP with secondary dystonia, aged between 3-15 years were included in the study.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
The Barry-Albright Dystonia Scale (BADS) | baseline
  The Barry-Albright Dystonia Scale designed for secondary dystonia and presence of dystonia in various body parts. It is a 5-point, criterion-based, ordinal scale designed to assess dystonia in eight body regions: eyes, mouth, neck, trunk, and the four extremities. Raters score dystonia as none (0), slight (1), mild (2), moderate (3), or severe (4).
The Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD) | baseline
  The Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD) is a measure of caregivers' perceptions of activity limitations, health status, well-being, and ease of care for children with severe cerebral palsy (CP). The CPCHILD consists of 36 items comprising the following domains: (1) Personal Care; (2) Positioning, Transfer, and Mobility; (3) Communication and Social Interaction; (4) Comfort, Emotions, and Behavior; (5) Health; and (6) Overall Quality Of Life.
The Care and Comfort Hypertonicity Questionnaire (CCHQ) | baseline
  The Care and Comfort Hypertonicity Questionnaire (CCHQ) is an interview questionnaire consisting of 27 questions divided into four scales: personal care,positioning/transferring, comfort and interaction/communication. Questions are answeredusing a 7-point Likert scale; mean scale score is calculated. The interview takes approximately10 min to administer. It provides a measure of functional limitation and has some quality-of-life elements with questions relating to pain and self-esteem. It indicates disease severity interms of degree of disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem Altunizade Hospital, Istanbul, Altunizade, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.